CLINICAL TRIAL: NCT04047056
Title: Analisys of the Effectiveness of Laboral Kinesiotherapy in Prevention of Upper Limb Musculoskeletal Disorders in the Workers of a University Hospital
Brief Title: Effectiveness of Laboral Kinesiotherapy in Prevention of Upper Limb Musculoskeletal Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Apoio ao Ensino, Pesquisa e Assistência do Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto da Universidade de São Paulo (Other); Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Marisa de Cassia Registro Fonseca, Clinical Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: FMRPUSP3
Record Dates: First submitted 2019-07-31; First posted 2019-08-06 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Upper Limb; Injury, Superficial, Multiple
Keywords: physiotherapy; prevention; pain; upper limb; exercises; musculoskeletal disorders
MeSH Terms: conditions — Wounds and Injuries; Pain; Motor Activity; Musculoskeletal Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ergonomic Guidelines Manual (Placebo Comparator): A manual of ergonomic occupational and daily living guidelines will be given to both control and labor kinesiotherapy groups, which is the only approach for the control group initially.
  Interventions: Other: Labor Kinesiotherapy
- Labor Kinesiotherapy in group (Active Comparator): The intervention will be performed by a physical therapist, which will consist of preparatory labor kinesiotherapy, which aims to prepare the workers' osteo-articular system for the beginning of the work activity, acting more specifically on those muscle groups that will be most required during the journey which will be identified in the evaluation. Labor kinesiotherapy will be performed in the workplace before the workday and will last 20 minutes, 3 times a week, for 12 weeks.
  Interventions: Other: Labor Kinesiotherapy

INTERVENTIONS:
Other: Labor Kinesiotherapy — The intervention group will perform 5 minutes of warm-up with free active exercises, 10 minutes of specific resistance exercises for the cervical and upper limbs and 5 minutes of stretching and muscle relaxation.The initial free active exercises will be performed in 3 sets of 15 repetitions; Resistance exercises will be performed in 3 sets of 10 repetitions and stretching will be performed in 3 sets of 30 seconds.
  Regarding the intervals between exercises, active recovery will be adopted to counteract the effects of muscle fatigue.

SUMMARY:
ABSTRACT

Work-related musculoskeletal disorders are seen as a public health problem, and can often lead to temporary or permanent incapacity to work. Exercises can be indicated to prevent musculoskeletal disorders, allied to ergonomic intervention as a preventive approach. Objectives: The objective of this study is to analyze the effects of workplace muscle strengthening kinesiotherapy in the reduction of pain and discomfort in the upper limbs and cervical region perceived by the workers of a university hospital. Methods: After a priori sample size calculation based on pain numeric scale, 166 volunterrs will be recruted and assigned randomly to the "labor kinesiotherapy" group (GCL) or to the "control group" (CG), considering 10% sample size lost and intention to treat. The primary outcomes will be the pain perceived by the Numerical Pain Scale (NDT) and Nordic Questionnaire, and isokinetic muscle strength through the mean peak torque work of shoulder abduction. The discomfort and disability will be evaluated by the PSFS and QuickDASH questionnaires. The Ergonomic Analysis of Work will be evaluated by the manual "Ergonomic Analysis Focused on Activities" - EAFA and application of QEC, RULA, REBA and HARM tools. Statistical analysis will be performed through PASW Statistics ™, version 20.0. The independent sample T test will be used to compare the groups. The Cohen index will be set for the effect size calculation. All analyzes will be conducted with 95% confidence interval and p <0.05 significance.

ELIGIBILITY:
Inclusion Criteria:

* Workers who have or do not have musculoskeletal complaints in the cervical, shoulder, elbow, wrist or hand and / or fingers, without clinical diagnosis and who are not away from their professional activities.

Exclusion Criteria:

* Workers presenting:

  * Pregnancy;
  * Congenital abnormality of the spine and significant musculoskeletal deformities (such as amputation, dysmetria);
  * Severe cervical spine disorders, postoperative conditions in the neck or upper limb region;
  * Uncontrolled cardiovascular disease, cardiac arrhythmia, angina or related symptoms, and postural hypotension or other contraindications to exercise;
  * Workers who engage in some form of regular physical activity involving muscle strengthening and endurance exercises.
  * Workers who have a proven diagnosis of upper limb musculoskeletal dysfunction and are undergoing physical therapy treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2023-01-25 (Actual)

PRIMARY OUTCOMES:
Numerical Pain Scale - NPS | 12 weeks.
  Difference in numerical pain scale in the 3 evaluations. The numerical pain scale score ranges from 0 to 10, with values closer to 10 indicating worse pain.
shoulder abduction Torque peak in the Isokinetic Dynamometer | 12 weeks.
  Mean difference in torque peak achieved by the Isokinetic Dynamometer at baseline and after 12 weeks.

SECONDARY OUTCOMES:
Quick Disabilities of de Arm, Shoulder and Hand (QuickDAS) | 12 weeks.
  Difference in DASH questionnaire scores in 3 evaluations. The QuickDASH score ranges from 0 to 100, with values closer to 100 indicating better health.
Patient Specific Functional Scale (PSFS) | 12 weeks.
  Difference in PSFS questionnaire scores in 3 evaluations. The PSFS allows patients to report on their functional status at baseline and at a follow-up session, to determine if a meaningful change in functional status has occurred.

CONTACTS AND LOCATIONS:
Locations (1):
- Natalia Claro da Silva, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] da Silva NC, Ricci FPFM, de Castro VR, de Lima ACR, do Carmo Lopes ER, de Salvo Mauad LD, Kawano Suzuki KA, de Oliveira Medeiros ME, de Santana JS, Rocha FLR, de Cassia Registro Fonseca M. Effects of workplace upper extremity resistance exercises on function and symptoms of workers at a tertiary hospital: a randomized controlled trial protocol. BMC Musculoskelet Disord. 2022 Feb 5;23(1):119. doi: 10.1186/s12891-022-05059-5. PMID 35123476